CLINICAL TRIAL: NCT05853471
Title: Evaluation of [18F]MC225-PET to Measure P-glycoprotein Function in Neurodegenerative Disease
Brief Title: [18F]MC225-PET in Neurodegenerative Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Gert Luurtsema, Principal Investigator, University Medical Center Groningen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202100647
Record Dates: First submitted 2022-11-09; First posted 2023-05-10 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Neurodegenerative Diseases; Alzheimer Disease; Parkinson Disease; Mild Cognitive Impairment
Keywords: PET; pharmacokinetic modeling; [18F]MC225
MeSH Terms: conditions — Neurodegenerative Diseases; Alzheimer Disease; Parkinson Disease; Cognitive Dysfunction | interventions — MC225 compound

STUDY DESIGN:
Intervention Model Description: [18F]MC225 is administrated to patients in three groups to evaluate the P-glycoprotein function in these groups and compare the results with the P-gp function of healthy volunteers obtained in a previous study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alzheimer's disease (Active Comparator): Patients diagnosed with Alzheimer's disease
  Interventions: Drug: [18F]MC225
- Mild Cognitive Impairment (Active Comparator): Patients diagnosed with Mild Cognitive Impairment
  Interventions: Drug: [18F]MC225
- Parkinson's disease (Active Comparator): Patients diagnosed with Parkinson's disease
  Interventions: Drug: [18F]MC225

INTERVENTIONS:
Drug: [18F]MC225 — All participants will undergo a PET scan with [18F]MC225. No pharmaceutical effects are expected and the study will exclusively have a diagnostic purpose. However, since [18F]MC225 is a new PET tracer, it is included in pharmaceutical studies and any study performed with [18F]MC225 will be automatically be registered as intervention study.

SUMMARY:
P-glycoprotein, an efflux transporter at the blood-brain barrier plays an important role in de development of neurodegenerative disease. A novel PET tracer ([18F]MC225) was developed to measure the function of P-glycoprotein and was tested with succes in healthy volunteers. This study aims to evaluate [18F]MC225 in neurodegenerative disease.

DETAILED DESCRIPTION:
A decrease in P-glycoprotein (P-gp) function is associated with the onset of neurodegenerative disease. New treatment strategies in neurodegenerative disease, including Parkinson's disease and Alzheimer's disease, aim to restore the P-gp function. To evaluate the effect of these potential therapies, measurement of the P-gp function is necessary. Up until now [11C]verapamil is considered to be the gold standard to measure P-gp function. However tracer uptake in the brain of [11C]verapamil is too low for adequate measurement of treatment effect, especially of restoring P-gp function. A novel PET tracer to measure P-gp function, [18F]MC225, has the potential advantage of higher brain uptake values at baseline and might therefore able to measure both up- and down regulation P-gp function. [18F]MC225 was recently studied in healthy volunteers and a method to quantify P-gp function was developed. This study aims to evaluate [18F]MC225 to measure P-gp function in neurodegenerative disease.

To this aim 10 MCI patients, 10 patients with Alzheimer's disease and 10 Parkinson's disease patients will be included and undergo one 60 min dynamic [18F]MC225 PET scan, combined with a 10 min [15O]H2O PET. Tracer uptake values (Vt) and influx (K1) in several brain regions of interest, representing local P-gp function will be compared with the [18F]MC225 uptake values in the brain of healthy volunteers obtained in a previous study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is diagnosed with Alzheimer's disease, Parkinson's disease or Mild Cognitive Impairment

Exclusion Criteria:

* Use of any medication influencing the P-glycoprotein function
* History of neuropsychiatric disorders
* Contra-indications MRI
* Allergy contrast agent

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
P-glycoprotein function | 60 minutes
  The function of P-glycoprotein at the blood-brain barrier measured by PET tracer-uptake (volume of distribution) in the brain

CONTACTS AND LOCATIONS:
Overall Officials: Gert Luurtsema, Phd, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers